CLINICAL TRIAL: NCT02697357
Title: Emotion Regulation Therapy to Address Distress Among Caregivers
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Hunter College of City University of New York (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 15-219
Record Dates: First submitted 2016-02-24; First posted 2016-03-03 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Care Givers
Keywords: Emotion Regulation Therapy; Distress Among Caregivers; 15-219

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — optional blood sample and a saliva sample

GROUPS / COHORTS (1):
- Caregivers: This study is a pilot, single-arm intervention of Emotion Regulation Therapy for Cancer Caregivers (ERT-C). We plan to recruit a pilot sample 32 consented (24 evaluable) caregivers of patients diagnosed with cancer and measure their distress, anxiety, and other psychological outcomes at baseline. Caregivers will be consented into an 8-session ERT-C therapy (approximately 12 - 16 weeks).
  Interventions: Behavioral: Psychosocial Instruments; Behavioral: Emotion Regulation Therapy for Cancer Caregivers (ERT-C)

INTERVENTIONS:
Behavioral: Psychosocial Instruments
Behavioral: Emotion Regulation Therapy for Cancer Caregivers (ERT-C)

SUMMARY:
The aim of this study is to adapt and pilot test a type of therapy called Emotion Regulation Therapy (ERT-C) for informal caregivers of patients with cancer. Informal caregivers include partners, family members, children, parents, and friends providing informal care to a patient. Providing care to someone with cancer can be difficult. The purpose of this intervention is to improve coping and physical well-being among caregivers, which in turn will allow them to provide better care for their loved ones. Investigators would also like to learn about biological factors like stress that may affect one's emotional and physical well-being. This study will allow to better understand caregivers needs, and further develop a program to provide services to caregivers within MSKCC community and nationwide.

ELIGIBILITY:
Inclusion Criteria:

* As per self-report, age 18 or over
* As per self-report, a current caregiver to a patient with any site or stage of cancer
* score of ≥ 4 on the Distress Thermometer (DT) and indication that this distress is related in some way to the caregiving role. Potential participants will be asked whether or not their distress is in any way related to their caregiving experience. Individuals who answer "no" will be asked whether or not their distress started or has gotten worse since the patient began treatment or was diagnosed.
* Either a score of ≥ 15 on the Brief Penn State Worry Questionnaire OR a score > 12 on the Brooding Subscale of the Rumination Response Scale
* In the judgment of the investigators and/or consenting professional, able to read and comprehend English
* In the judgment of the consenting professional cognitively able to provide informed consent

Exclusion Criteria:

* As per self-report, a lifetime history of bipolar disorder, schizophrenia, or schizoaffective disorder
* In the judgment of the consenting professional is unable to provide informed consent and complete study sessions and assessment.
* If participating in optional biospecimen collection;as per self-report, has medical conditions that affect the immune system and would confound immune evaluation (e.g., autoimmune disorder, inflammatory disease; uncontrolled thyroid disease; active infection; myocardial infarction or stroke in the last 6 months; Type I diabetes; acute hepatitis; recent vaccination for viral disease)
* As per self-report, is a regular smoker (daily use)
* As per self-report, is a heavy drinker (regularly having more than 14 alcoholic beverages per week for men, 7 for women)
* As per self- report, engaging in night shift work
* As per self- report, currently engaged in ongoing psychotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from outpatient clinics in various departments at MSKCC, including the Department of Psychiatry & Behavioral Sciences, Social Work, Neurology, Integrative Medicine and Bone Marrow Transplant services.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
number of patients completing at least 6 out of the 8-sessions | 1 year
  feedback from participants by qualitative research methods

CONTACTS AND LOCATIONS:
Overall Officials: Allison Applebaum, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/